CLINICAL TRIAL: NCT07035197
Title: Facilitators and Barriers to Eptinezumab Administration in Thailand: Real-World Experiences and Perspectives From Mixed-method Design and In-Depth Interviews (FACEpi)
Brief Title: Facilitators and Barriers to Eptinezumab Administration in Thailand
Acronym: FACEpi
Status: Recruiting | Type: Observational
Sponsor: Chulalongkorn University (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Thanakit Pongpitakmetha, MD, MSc, Lecturer, Chulalongkorn University
Other Study IDs: Med Chula IRB 0329/68
Record Dates: First submitted 2025-06-03; First posted 2025-06-25 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-06

CONDITIONS: Migraine; Treatment; Treatment Refusal
Keywords: Migraine; CGRP; Eptinezumab; Mixed method; Real world; Thailand; Treatment; Barrier; Facilitator; Interview
MeSH Terms: conditions — Migraine Disorders; Treatment Refusal | interventions — eptinezumab; salicylhydroxamic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- People with episodic or chronic migraine who have NEVER received CGRP mAb therapy: Patients who were diagnosed migraine with or without aura or chronic migraine and have NEVER received eptinezumab.
  Inclusion
  1. Age ≥ 18 years
  2. Diagnosed with migraine with or without aura or chronic migraine according to the ICHD-3
  3. Have received eptinezumab infusion at KCMH
  4. Have NEVER received any CGRP mAbs prior to starting eptinezumab
  5. Able to communicate in Thai fluently
  6. Provide informed consent
  Exclusion
  1. Participants who cannot completely participate in an in-depth interview and questionnaires, either in-person or online
  2. Participants with headache disorders other than migraine with or without aura or chronic migraine
  3. Alcohol or drug use that, in the opinion of the investigator, would interfere with completion of study procedures
  4. A known history of allergy to eptinezumab
  Interventions: Drug: Eptinezumab
- People with episodic or chronic migraine who have received CGRP mAb therapy: Patients who were diagnosed migraine with or without aura or chronic migraine and have received eptinezumab.
  Inclusion
  1. Age ≥ 18 years
  2. Diagnosed with migraine with or without aura or chronic migraine according to the ICHD-3
  3. Have received eptinezumab infusion at the KCMH
  4. Have received other CGRP mAbs prior to starting eptinezumab
  5. Able to communicate in Thai fluently
  6. Provide informed consent
  Exclusion
  1. Participants who cannot completely participate in an in-depth interview (IDI) and questionnaires, either in-person or online
  2. Participants with headache disorders other than migraine with or without aura or chronic migraine
  3. Alcohol or drug use that, in the opinion of the investigator, would interfere with completion of study procedures
  4. A known history of allergy to eptinezumab
  Interventions: Drug: Eptinezumab
- Healthcare Provider: Healthcare providers (e.g. doctor, outpatient nurse and daycare nurse) who are responsible for providing eptinezumab to the patients.
  Inclusion criteria
  1. Age ≥ 18 years
  2. Currently working at KCMH
  3. Have been working at KCMH for more than 3 months
  4. Involved in providing care to patients attending the Headache Clinic
  5. Able to communicate in Thai fluently
  6. Provide informed consent
  Exclusion criteria
  1. Participants who cannot completely participate in an IDI, either in-person or online
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Drug: Eptinezumab — Eptinezumab 100 mg IV q 3 months
  * Baseline visit: Within 24 hours of receiving eptinezumab (duration of IDI ~30 - 45 minutes)
    * Semi-structured In-depth interview
    * MMD (days)
    * Thai version MIDAS (total score, grading)
    * Thai version EQ-5D-5L (5 domains & 5 levels of severity; index score)
  * 3-month follow-up visits (duration of interview: ~10 minutes):
    * Semi-structured brief interview
    * MMD (days)
    * Thai version MIDAS (total score, grading)
    * Thai version EQ-5D-5L (5 domains & 5 levels of severity; index score)
  * 6-month follow-up visit:
    * no interview
    * MMD (days)
    * Thai version MIDAS (total score, grading)
    * Thai version EQ-5D-5L (5 domains & 5 levels of severity; index score)
  Groups: People with episodic or chronic migraine who have NEVER received CGRP mAb therapy; People with episodic or chronic migraine who have received CGRP mAb therapy
Other: Sham (No Treatment) — ** No intervention, neither eptinezumab nor placebo, was given
  * Baseline visits: Within 24 hours of giving eptinezumab administration (duration of IDI ~30 - 45 minutes) - Semi-structured in-depth interview
  Groups: Healthcare Provider

SUMMARY:
This research study is designed as a longitudinal prospective descriptive study using mixed-method data collection. Eptinezumab, an anti-calcitonin gene-related peptide monoclonal antibody (anti-CGRP mAb), is administered by intravenous (IV) infusion every 3 months as preventive medication for individuals with migraine who have been diagnosed based on theInternational Classification of Headache Disorders, 3rd edition (ICHD-3) by headache specialist neurologists. The goal of this study is to understand the real-life experiences of people with migraine who receive eptinezumab in a hospital setting in Thailand, a middle-income country. The researchers want to learn about what makes it easier or harder for patients and healthcare workers to use this treatment.

The main questions it aims to answer are:

* What are the barriers and facilitators to using eptinezumab from the perspectives of patients and healthcare providers?
* Does eptinezumab reduce monthly migraine days and improve quality of life over time?

Participants will:

* (For migraine patients) Take part in an in-depth interview (IDI) within 24 hours after receiving an eptinezumab infusion
* (For migraine patients) Complete questionnaires about migraine symptoms, disability, and quality of life at baseline, 3 months, and 6 months
* (For healthcare providers) Take part in a one-time interview about their experiences administering eptinezumab

The study will also look at how well eptinezumab works by measuring changes in monthly migraine days and other health scores over a 6-month period. The information from this study may help improve migraine care in Thailand and support better access to new treatments like eptinezumab.

DETAILED DESCRIPTION:
This study explores how people with migraine in Thailand experience treatment with eptinezumab, a anti-CGRP mAb given through an IV infusion every 12 weeks to help prevent migraine attacks. While this medicine may work quickly and avoid skin irritation from injections, it must be given at a hospital, which may cause challenges for patients and healthcare providers. These challenges can include travel, time, cost, or extra work for hospital staff.

The study, called FACEpi, will look at what makes eptinezumab easy or hard to use in real life. It will gather views from both people with migraine and the healthcare professionals who provide the treatment. Researchers want to better understand how patients feel about this treatment and how it affects their daily life.

About 30 participants will join the study from the Headache Clinic and Daycare Ward at King Chulalongkorn Memorial Hospital (KCMH). These include adults with migraine (10 participants who have never recieved anti-CGRP mAb and 10 participants who have recieved anti-CGRP mAb) and 10 healthcare providers including doctors, nurses, nurse aids, etc. who give eptinezumab in our hospital.

Each patient will take part in a semi-structured interview shortly after receiving eptinezumab and complete short surveys about migraine symptoms, migraine headache day (MHD), migraine disability (MIDAS), and quality of life (Euro-Quality of Life version EQ-5D-5L) at three time points: within 24 hours after treatment, after 3 months, and after 6 months. Healthcare providers will complete a one-time interview to talk about their experiences giving the treatment.

The main goals of this study are:

* To understand what helps or makes it hard to use eptinezumab in real-world practice
* To see if eptinezumab helps reduce migraine days and improve quality of life

Data from interviews will be reviewed for common themes using special software. Outcome measures will be analyzed using standard statistical tools. The results of this study will help doctors and public health leaders understand how to make migraine treatment more accessible and effective for patients in Thailand.

ELIGIBILITY:
Target Population

* Group 1: Patients who were diagnosed migraine with or without aura or chronic migraine and have received eptinezumab.
* Group 2: Healthcare providers (e.g. doctor, outpatient nurse and daycare nurse) who are responsible for providing eptinezumab to the patients.
* Inclusion Criteria Group 1: People with migraine with or without aura or chronic migraine Inclusion criteria Group 1A

  1. Age ≥ 18 years
  2. Diagnosed with migraine with or without aura or chronic migraine according to the International Classification of Headache Disorders, 3rd edition (ICHD-3)*
  3. Have received eptinezumab infusion at the King Chulalongkorn Memorial Hospital (KCMH)
  4. Have received other CGRP mAbs prior to starting eptinezumab
  5. Able to communicate in Thai fluently
  6. Provide informed consent Group 1B

  <!-- -->

  1. Age ≥ 18 years
  2. Diagnosed with migraine with or without aura or chronic migraine according to the ICHD-3*
  3. Have received eptinezumab infusion at the KCMH
  4. Have NEVER received any CGRP mAbs prior to starting eptinezumab
  5. Able to communicate in Thai fluently
  6. Provide informed consent

     * The diagnosis will be established by consensus between two headache specialists. In case of a discrepancy, conflicts will be resolved through a final consensus agreement between the two specialists prior to enrollment.

     Group 2: Healthcare providers Inclusion criteria

  <!-- -->

  1. Age ≥ 18 years
  2. Currently working at KCMH
  3. Have been working at KCMH for more than 3 months
  4. Involved in providing care to patients attending the Headache Clinic
  5. Able to communicate in Thai fluently
  6. Provide informed consent
* Exclusion Criteria Group 1: People with migraine with or without aura or chronic migraine

  1. Participants who cannot completely participate in an in-depth interview (IDI) and questionnaires, either in-person or online
  2. Participants with headache disorders other than migraine with or without aura or chronic migraine
  3. Alcohol or drug use that, in the opinion of the investigator, would interfere with completion of study procedures
  4. A known history of allergy to eptinezumab Group 2: Healthcare providers

  <!-- -->

  1. Participants who cannot completely participate in an IDI, either in-person or online

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Group 1: Patients who were diagnosed migraine with or without aura or chronic migraine and have received eptinezumab.
  * Group 2: Healthcare providers (e.g. doctor, outpatient nurse and daycare nurse) who are responsible for providing eptinezumab to the patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Migraine patients' experiences after receiving eptinezumab | At enrollment (witihin 24 hours of receiving eptinezumab) and 3 months follow-up
  Group 1 (People with migraine with or without aura or chronic migraine):
  1. Baseline visit at the time of enrollment.
     - A semi-structured IDI will be conducted within 24 hours of receiving eptinezumab.
  2. 3-month follow-up visit:
     * Participants will complete a set of questionnaires to assess their experiences after receiving eptinezumab infusion
     * A brief semi-structure interview
  3. 6-month follow-up visit:
     * No interview
Facilitators and barriers of integrating the use of eptinezumab in the headache specialty clinic in Thailand from the perspective of migraine patients | At enrollment (witihin 24 hours of receiving eptinezumab) and 3 months follow-up
  Group 1 (People with migraine with or without aura or chronic migraine)
  * Baseline visit: Within 24 hours of receiving eptinezumab
    - Semi-structured IDI (duration of IDI ~30 - 45 minutes)
    * Satisfactory, acceptance, adaptability, feasibility, cost of eptinezumab administration
    * Patients' migraine symptoms and their impact on daily life, emotional well-being, and social well-being.
    * The perspective of oral and non-oral form of prevention medicine
    * Patients' experiences of migraine symptom improvement and the wearing-off effect during prior anti-CGRP injections in the group with previously failed anti-CGRP treatments.
    * Patients' migraine symptoms between administration of eptinezumab
  * 3-month follow-up visits (duration of interview: ~10 minutes)
    * Brief interview (duration of interview: ~10 minutes)
      * What are your thoughts on eptinezumab infusion?
      * What is the difference between prior anti-CGRP treatments and eptinezumab in prior anti CGRP group?
Facilitators and barriers of integrating the use of eptinezumab in the headache specialty clinic in Thailand from the perspective of healthcare providers | At enrollment (witihin 24 hours of giving eptinezumab administration)
  Group 2 (Healthcare providers) o Baseline visits: Within 24 hours of giving eptinezumab administration (duration of IDI ~30 - 45 minutes)
  - Semi-structured IDI exploring facilitators and barriers of integrating the use of eptinezumab in the headache specialty clinic in Thailand

SECONDARY OUTCOMES:
Changes in monthly migraine days (MMD) | At enrollment (witihin 24 hours of receiving eptinezumab), 3 months follow-up, and 6 months follow-up
  Group 1 (People with migraine with or without aura or chronic migraine)
  Monthly migraine days are measured by patient self-report or headache diary review by investigators.
Changes in Migraine Disability Assessment (MIDAS) Score | At enrollment (witihin 24 hours of receiving eptinezumab), 3 months follow-up, and 6 months follow-up
  The MIDAS score is a validated questionnaire used to quantify migraine-related disability over the past 3 months. It consists of five main items assessing the number of days of activity limitation due to migraine in three domains: work/school, household chores, and social/leisure activities.
  Scoring The total MIDAS score (Minimum value: 0 Maximum value: 270 Higher scores mean a worse disability) is calculated by summing responses to the five main items (each answered as the number of days affected).
  Disability Severity Grading:
  * Grade I (0-5): Little or no disability
  * Grade II (6-10): Mild disability
  * Grade III (11-20): Moderate disability
  * Grade IV (21+): Severe disability
  Two additional questions assess number of headache days per 3 months and average headache pain intensity (on a scale of 0-10), but these do not contribute to the total score.
  Thai MIDAS version was applied and administered by trained investigators https://doi.org/10.31524/bkkmedj.2018.02.003
Changes in Quality of Life (EuroQoL (EQ-5D-3L)) | At enrollment (witihin 24 hours of receiving eptinezumab), 3 months follow-up, and 6 months follow-up
  Quality of life as measured by the Thai version of the EQ-5D-5L questionnaire. The raw scores were transformed to utility scores for Thai population as previously suggested (Pattanaphesaj J., 2018).
  Structure The EQ-5D-3L includes:
  * Five dimensions:
    1. Mobility
    2. Self-care
    3. Usual activities
    4. Pain/discomfort
    5. Anxiety/depression Each dimension has three levels:
  * No problems (Level 1)
  * Some problems (Level 2)
  * Extreme problems (Level 3) The combination of levels across dimensions defines a unique health state (e.g., 11223). A total of 243 health states are possible.
  Scoring
  * Each health state is converted into a single index value (utility score) using a Thai-specific value set.
  * Utility scores typically range from -0.452 to 1.000, where:
  * 1.000 = full health
  * 0 = death
  * <0 = states perceived worse than death
Changes in abortive medication use | At enrollment (witihin 24 hours of receiving eptinezumab), 3 months follow-up, and 6 months follow-up
  Abortive medication use is reviewed by patient self-report and rechecked with the electronic medical record information by investigators
  Data collection
  * Generic name
  * Dosage (mg)
  * Number of pills used per month
Change in preventive medication use | At enrollment (witihin 24 hours of receiving eptinezumab), 3 months follow-up, and 6 months follow-up
  Preventive medication use is reviewed by patient self-report and rechecked with the electronic medical record information by investigators
  Data collection
  * Generic name
  * Dosage (mg)
  * Number of pills used per month

CONTACTS AND LOCATIONS:
Overall Officials: Prakit Anukoolwittaya, MD, Principal Investigator — Division of Neurology, Department of Medicine, King Chulalongkorn Memorial Hospital, The Thai Red Cross Society; Thanakit Pongpitakmetha, MD, MSc, Study Director — Department of Pharmacology, Faculty of Medicine, Chulalongkorn University; Sekh Thanprasertsuk, MD, Study Director — Department of Physiology, Faculty of Medicine, Chulalongkorn University; Akarin Hiransuthikul, MD, MSc, Study Director — Department of Preventive and Social Medicine, Faculty of Medicine, Chulalongkorn University; Wanakorn Rattanawong, MD, Study Director — Faculty of Medicine, King Mongkut's Institute of Technology Ladkrabang
Locations (1):
- King Chualongkorn Memorial Hospital, the Thai Red Cross Society, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Argoff C, Herzog SP, Smith RM, Kotak SV, Sopina L, Saltarska Y, Soni-Brahmbhatt S, Khan FA. Real-world effectiveness and satisfaction with intravenous eptinezumab treatment in patients with chronic migraine: REVIEW, an observational, multi-site, US-based study. J Headache Pain. 2024 Apr 25;25(1):65. doi: 10.1186/s10194-024-01764-9. PMID 38664605
- [Background] Zhao YJ, Ong JJY, Sonu SK, Dang J, Ng CC, Herr KJ, Bose R, Jion YI. A real-world prospective observational study of eptinezumab in Asian patients with migraine. Headache. 2024 Jul-Aug;64(7):810-824. doi: 10.1111/head.14737. Epub 2024 May 24. PMID 38785386
- [Background] Winner PK, McAllister P, Chakhava G, Ailani J, Ettrup A, Krog Josiassen M, Lindsten A, Mehta L, Cady R. Effects of Intravenous Eptinezumab vs Placebo on Headache Pain and Most Bothersome Symptom When Initiated During a Migraine Attack: A Randomized Clinical Trial. JAMA. 2021 Jun 15;325(23):2348-2356. doi: 10.1001/jama.2021.7665. PMID 34128999
- See also: Thai version of the Migraine Disability Assessment Score (MIDAS) — https://he02.tci-thaijo.org/index.php/bkkmedj/article/view/222195